CLINICAL TRIAL: NCT06083441
Title: SeeMe: A Pilot Study Developing Predictive, Real-Time Consciousness Assessment Metrics Based on Facial Expression Changes
Brief Title: SeeMe: An Automated Tool to Detect Early Recovery After Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Sima Mofakham, Assistant Professor and Director of Research, Stony Brook University
Other Study IDs: IRB2019-00199
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Disorder of Consciousness; Consciousness, Loss of; Trauma, Brain; Traumatic Brain Injury; Acute Brain Injury
Keywords: Consciousness; Acute brain injury; Consciousness Recovery; Consciousness Measurement; Facial Motion Analysis; Microscopic movements; Traumatic Brain Injury
MeSH Terms: conditions — Consciousness Disorders; Unconsciousness; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acute Brain Injury (ABI): Patients that have suffered an ABI resulting in Coma (Glasgow Coma Scale (GCS) < 9) will undergo SeeMe and CRS-R assessment once a day until hospital discharge
  Interventions: Diagnostic Test: SeeMe; Diagnostic Test: Coma Recovery Scale-Revised (CRS-R)
- Control: Healthy subjects will undergo SeeMe and CRS-R assessment once.
  Interventions: Diagnostic Test: SeeMe; Diagnostic Test: Coma Recovery Scale-Revised (CRS-R)

INTERVENTIONS:
Diagnostic Test: SeeMe — A video-recorded SeeMe command following assessment by a trained professional once a day Each session involves three command sets that are played from an audio recording 10 times over the course of 8 minutes. These commands are "Stick out your tongue", "Open your eyes", and "Show me a smile" Each command set is recorded separately for a total of 3 videos per session. These videos are then analyzed by SeeMe to detect if subjects are responding to commands.
  Other Names: SeeMe session
Diagnostic Test: Coma Recovery Scale-Revised (CRS-R) — A video-recorded CRS-R score assessment by a trained professional once a day. A score of 10 or greater, an auditory score >2, or an arousal score > 0 means that a subject is responding to commands

SUMMARY:
Early prediction of outcomes after acute brain injury (ABI) remains a major unsolved problem. Presently, physicians make predictions using clinical examination, traditional scoring systems, and statistical models. In this study, we will use a novel technique, "SeeMe," to objectively assess the level of consciousness in patients suffering from comas following ABI. SeeMe is a program that quantifies total facial motion over time and compares the response after a spoken command (i.e. "open your eyes") to a pre-stimulus baseline.

DETAILED DESCRIPTION:
Acute brain injury (ABI) recovers at a variable rate. While some progress has been made in predicting long-term outcomes in traumatic brain injury (TBI) and intracranial hemorrhage, there is a critical need for short-term prediction of outcomes, in the first days and weeks after injury. With advances in machine learning and artificial intelligence, there is a growing interest in facial analysis and its application in neurological and psychiatric disorders. Here we describe "SeeMe," a novel automated objective measure of consciousness based on microexpression analyses in response to auditory commands. In measuring the smallest muscular movements undetectable by clinical observation, this technique has the high spatial resolution needed to detect hidden signs of recovery and the high temporal resolution needed to study neural circuits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Healthy Volunteers
* Comatose patients (patients with a GCS < 9) due to an acute brain injury (traumatic brain injury, spontaneous subarachnoid hemorrhage, severe meningoencephalitis, etc.)

Exclusion Criteria:

* A history of a neurologically debilitating disease (i.e., dementia, glioblastoma, Alzheimer's, multiple sclerosis, major vessel stroke, previous severe TBI, etc.)
* Any other medical condition that, in the judgment of the investigator, makes participation in the study unsafe.
* Pregnant subjects
* Comatose patients without a legal authorized representative (LAR)
* Prisoners or wards of the state
* Persons who have not attained the legal age for consent to treatments or procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers: Adults 18-85 years old with no history of a neurologically debilitating disease (i.e., dementia, glioblastoma, Alzheimer's, multiple sclerosis, major vessel stroke, previous severe TBI, etc.) that are recruited via flyer and word of mouth
  Patients in a coma: Adults 18-85 years old with no history of a neurologically debilitating disease that are comatose (GCS < 9) due to an acute brain injury. Patients in a comatose state will be identified during neurosurgical consultation in the hospital by the study physicians
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Detection of Command Following | Measured Daily from enrollment until subject is following commands or date of death of any cause, whichever comes first, up to 60 days.
  Length of time until an intervention is able to detect that a subject is following commands

CONTACTS AND LOCATIONS:
Overall Officials: Sima Mofakham, PhD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng F, Yu J, Xiong H. Facial expression recognition in JAFFE dataset based on Gaussian process classification. IEEE Trans Neural Netw. 2010 Oct;21(10):1685-90. doi: 10.1109/TNN.2010.2064176. Epub 2010 Aug 19. PMID 20729164
- [Background] Zhao Y, Xu J. A Convolutional Neural Network for Compound Micro-Expression Recognition. Sensors (Basel). 2019 Dec 16;19(24):5553. doi: 10.3390/s19245553. PMID 31888182
- [Background] Valstar MF, Pantic M. Fully automatic recognition of the temporal phases of facial actions. IEEE Trans Syst Man Cybern B Cybern. 2012 Feb;42(1):28-43. doi: 10.1109/TSMCB.2011.2163710. Epub 2011 Sep 15. PMID 21926026
- [Background] Chouinard B, Scott K, Cusack R. Using automatic face analysis to score infant behaviour from video collected online. Infant Behav Dev. 2019 Feb;54:1-12. doi: 10.1016/j.infbeh.2018.11.004. Epub 2018 Nov 30. PMID 30508782
- [Background] Saadon JR, Yang F, Burgert R, Mohammad S, Gammel T, Sepe M, Rafailovich M, Mikell CB, Polak P, Mofakham S. Real-time emotion detection by quantitative facial motion analysis. PLoS One. 2023 Mar 10;18(3):e0282730. doi: 10.1371/journal.pone.0282730. eCollection 2023. PMID 36897921
- [Background] Kalmar K, Giacino JT. The JFK Coma Recovery Scale--Revised. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):454-60. doi: 10.1080/09602010443000425. PMID 16350986